CLINICAL TRIAL: NCT06276712
Title: A Randomized Controlled Trial Comparing Titanium Grade V (KS) Versus Titanium Grade IV (TS) Implants for the Treatment of Edentulous Mandible
Brief Title: RCT Comparing KS Versus TS for Ovedenture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Assistent Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_5
Record Dates: First submitted 2023-04-24; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant; Dental Implant-Abutment Design; Edentulous Jaw
Keywords: Dental Implant; Overdenture; Implant-abutment connection
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: A multicenters, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: A blinded (when possible) outcome assessor will evaluate all the outcomes and will take the radiogram for centralized analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ks dental implant (Experimental): Implant placement in edentulous jaws for a prosthetic implant rehabilitation with implant-retained overdenture (mucosally supported), on two implants using KS implant with 3.5 mm of diameter
  Interventions: Device: Implant placement with 3.5 mm diameter KS implants.
- TS dental implant (Active Comparator): Implant placement in edentulous jaws for a prosthetic implant rehabilitation with implant-retained overdenture (mucosally supported), on two implants using TS implant with 3.5 mm of diameter
  Interventions: Device: Implant placement with 3.5 mm diameter TS implants.

INTERVENTIONS:
Device: Implant placement with 3.5 mm diameter KS implants. — Implant placement in edentulous jaws for a prosthetic implant rehabilitation with implant-retained overdenture (mucosally supported), on two implants. with 3.5 mm diameter KS implants.After osseointegration, both dental implants will receive definitive prosthesis.
  Arms: Ks dental implant
Device: Implant placement with 3.5 mm diameter TS implants. — Implant placement in edentulous jaws for a prosthetic implant rehabilitation with implant-retained overdenture (mucosally supported), on two implants. with 3.5 mm diameter TS implants.After osseointegration, both dental implants will receive definitive prosthesis.
  Arms: TS dental implant

SUMMARY:
To evaluate the clinical and radiographic outcomes of KS implants used to rehabilitate edentulous mandible with dental-retained overdentures, and to compare it with same treatment on TS implants

ELIGIBILITY:
Inclusion Criteria:

* Any edentulous patient (post-extractive sites must to be healed from at least 3 months), with sufficient bone height and width in the anterior mandible (between canines) to allow the placement of two implants of 3.5 mm diameter of at least 8.5 mm of length.
* 18 years or older, and able to sign an informed consent.
* Smokers will be included and categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day).
* In case of post-extractive sites, they must have been healing for at least 3 months before being treated in the study.

Exclusion Criteria:

Exclusion criteria

* General contraindications to implant surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Previous guided bone reconstruction at the intended implant sites.
* Uncontrolled diabetes.
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of implant failure | Up to 5 years
  Defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable.
Number of prosthesis failure | Up to 5 years
  Whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reaso
Number of complications | Up to 5 years
  echnical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, suppuration, peri-implantitis, etc.) complications will be considered.
Rate of implant stability | Up to 5 years
  The stability of each individual implant will be measured by the local blinded outcome assessors manually tightening the screws with a torque of 30 Ncm at abutment connection at initial loading. At 1,3 and 5 years after loading, individual implants will be manually tested for stability. Once the single crowns will be screwed, their stability will be assessed by rocking the crown with the handles of two dental instruments.

SECONDARY OUTCOMES:
Peri-implant marginal bone level changes | At 1,3 and 5 years
  Peri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured.
Patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  1. Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2. Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3. Would you undergo the same therapy again? Possible answers: "yes" or "no".